CLINICAL TRIAL: NCT03522038
Title: Functional Assessment-guided Angioplasty in Patients With Coronary Chronic Total Occlusion (FAGA-CTO)
Brief Title: Functional Assessment-guided Angioplasty in Patients With Coronary Chronic Total Occlusion
Acronym: FAGA-CTO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-CV-201801
Record Dates: First submitted 2018-04-11; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Coronary Occlusion; Angioplasty, Balloon, Coronary
Keywords: coronary chronic total occlusion; functional evaluation
MeSH Terms: conditions — Coronary Occlusion | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 samples of EDTA blood (2ml glass) and 1 sample of serum (5ml glass) will be retained in a biobank.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: percutaneous coronary intervention — PCI was performed using standard techniques. Antiplatelet and antithrombotic agents were prescribed according to current PCI guidelines. A procedure was considered successful when achieving TIMI flow grade 3 with <30% angiographic residual stenosis in the CTO vessel. All patients received drug-eluting stents and were discharged on dual antiplatelet therapy with duration of at least on year.

SUMMARY:
The aim of this study is to investigate the role of functional evaluation for predicting clinical outcome in patients with coronary chronic total occlusion (CTO) undergoing percutaneous coronary intervention (PCI), and to evaluate the clinical evidence for the using of fractional flow reserve (FFR), coronary flow reserve (CFR), index of myocardial resistance (IMR) and dynamic single photon emission computed tomography (D-SPECT) in these patients.

DETAILED DESCRIPTION:
PCI for CTO has dramatically changed in recent years. Although, with the improvement of devices and refinement of operator techniques, PCI of CTO can currently be performed with high success and low complication rates at experienced centers, the clinical benefit of recanalization of CTO is still a matter of debate. Accumulating evidence suggests that the improvement of left ventricular functional and prognosis is closely related with the area of viable myocardium, which has the potential for contractile recovery after revascularization. For the majority of interventional cardiologists, coronary angiography is the only invasive test deemed necessary for clinical decision-making, despite its weak ability to predict the functional impact of vascular occlusion on the subtended myocardium. To overcome this limitation, adjunctive diagnostic tools for functional evaluation, such as FFR, CFR, IMR and D-SPECT, have been introduced. In non-CTO patients, physiology-guided revascularization strategy has been definitely proven to be better than angiography-guided strategy in pivotal landmark studies. However, the clinical value of these functional parameters for the PCI of CTO is still unknown.

The aim of this study was to determine whether functional evaluation is a better predictor of clinical outcome in patients with CTO undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤80
* Patients diagnosed with CTO by coronary angiography
* Patient planned to receive PCI
* Diameter of CTO vessel > 2.25 mm

Exclusion Criteria:

* Age >80 or <18
* Myocardial infarction with 1 months
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary CTOs were defined as coronary lesions with Thrombolysis in Myocardial Infarction (TIMI) grade 0 flow of at least 3-month duration. Estimation of the occlusion duration was based on first onset of anginal symptoms, prior history of MI in the target vessel territory, or comparison with a prior angiogram.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline FFR at 6 months after CTO PCI | At baseline and 6 months after CTO PCI
  FFR measurement in donor vessels at were performed simultaneously using pressure wires (Abbot) before attempting the CTO vessel. FFR measurement in the CTO vessels were performed after the wire arrived at the distal true lumen through antegrade or retrograde route. The FFR in donor and CTO vessels were measured again after successful stenting of CTO vessels.
Change from Baseline FFR at 6 months after CTO PCI | At baseline and 6 months after CTO PCI
  CFR measurement in donor vessels at were performed simultaneously using pressure wires (Abbot) before attempting the CTO vessel. CFR measurement in the CTO vessels were performed after the wire arrived at the distal true lumen through antegrade or retrograde route. The CFR in donor and CTO vessels were measured again after successful stenting of CTO vessels.
Change from Baseline Myocardial perfusion at 6 months after CTO PCI | At baseline and 6 months after CTO PCI
  The myocardial perfusion before and after CTO PCI was evaluated by dynamic SPECT.
Change from Baseline Myocardial Viability at 6 months after CTO PCI | At baseline and 6 months after CTO PCI
  The myocardial viability before and after CTO PCI was evaluated by PET-MRI.

SECONDARY OUTCOMES:
MACE | 6 months after CTO PCI
  A major adverse cardiac event (MACE) was defined as the occurrence of cardiac death, nonfatal MI, and target lesion revascularization during the follow-up period.
In-stent restenosis | 6 months after CTO PCI
  In-stent restenosis was defined as >50% diameter stenosis by quantitative coronary angiography within a previously stented CTO vessel segment.

IPD SHARING:
Plan to Share IPD: No